CLINICAL TRIAL: NCT02371889
Title: A Randomized, Double-blind Placebo-Controlled Pharmacogenetic Study of Topiramate in European-American Heavy Drinkers
Acronym: TOPG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 821035; 821035 (Other: University of Pennsylvania); R01AA023192 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-02-26 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Alcoholism; Alcohol Use Disorder (AUD)
Keywords: Topiramate; Pharmacogenetics; Personalized Medicine
MeSH Terms: conditions — Alcoholism | interventions — Topiramate; Practice Management, Medical

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate + Medical Management (Experimental): Topiramate 200 mg/day orally in two divided doses. Dose will be titrated upward over a six-week period, maintained for 6 weeks, then tapered over 6 days + Medical Management sessions for 15-25 minutes per study visit
  Interventions: Drug: Topiramate; Behavioral: Medical Management
- Placebo Pill + Medical Management (Placebo Comparator): Inactive placebo with dosing schedule matched to intervention group + Medical Management sessions for 15-25 minutes per study visit
  Interventions: Behavioral: Medical Management; Drug: Inactive Placebo

INTERVENTIONS:
Drug: Topiramate — Max therapeutic dose of 200mg/day
  Other Names: Topamax
  Arms: Topiramate + Medical Management
Behavioral: Medical Management — Medical Management (MM; Pettinati, 2004) will support subjects' efforts to reduce or stop their drinking. The study nurse makes direct recommendations for reducing drinking to sensible levels. The first session will use the brochure A Guide to Sensible Drinking (WHO 1996). The subject is provided with information about pharmacotherapy and the importance of adherence to topiramate/placebo. Subsequent treatment sessions (15-25 minutes) will be conducted at each study visit, during which the nurse will perform an assessment of the subject's drinking, monitor his/her medication adherence, and make recommendations to follow until the next visit. Men will be advised to consume no more than 3 drinks 4 times per week; women will be advised to consume no more than 2 drinks 4 times per week.
  Other Names: MM
Drug: Inactive Placebo — In capsules indistinguishable from topiramate capsules and gradually increased to a maximum equivalent of 200 mg of topiramate/day
  Arms: Placebo Pill + Medical Management

SUMMARY:
The purpose of this study is to advance the effort to develop personalized pharmacotherapy for alcohol use disorders (AUDs). The investigators propose to conduct a 12-week, prospective, randomized clinical trial of the moderating effect of rs2832407 on the efficacy of TOP in reducing heavy drinking (HD) in 200 individuals of European descent with DSM-5 AUD. The investigators will stratify the randomization on genotype and oversample rs2832407*C homozygotes, the most TOP-responsive genotype, to ensure comparable numbers of patients in the four medication x genotype groups. The investigators will use daily data collection to examine changes in relevant process variables (e.g., alcohol expectancies) and their interaction with genotype and medication group as predictors of HD. The proposed study is innovative in that it will be the first prospective test of a pharmacogenetic hypothesis involving TOP; it will use daily reports to examine expectancies and how they interact with medication and genotype to predict HD; and it will enroll DSM-5 AUD patients whose goal is either to reduce or stop drinking, which will increase the study's external validity.

DETAILED DESCRIPTION:
This is a 12-week, prospective, randomized clinical trial of the moderating effect of rs2832407 on the efficacy of topiramate in reducing HD in 200 individuals of European descent with DSM-5 AUD. The investigators will stratify the randomization on genotype and oversample rs2832407*C homozygotes, the most topiramate-responsive genotype, to ensure comparable numbers of subjects in the four medication x genotype groups. The investigators will compare the efficacy of topiramate to placebo in reducing the frequency of HDDs in subjects with AUD using a two-arm, parallel-groups design. Subjects will either have a goal of reducing their drinking to safe levels or abstinence.

The investigators will use daily data collection to examine changes in relevant process variables and their interaction with genotype and medication group as predictors of HD. At each visit, all subjects will receive Medication Management (Pettinati, Weiss et al. 2004), which was developed for the COMBINE Trial and which the investigators modified to be relevant for both reducing heavy drinking and promoting abstinence. Random assignment to treatment group and double-blind conditions will be maintained throughout the study. Raters will be trained in the reliable use of all assessments. The investigators will use serum GGTP and percent disialotransferrin (%dCDT), an improved assay for carbohydrate deficient transferrin, to validate subject reports. Following a one-week pre-treatment assessment period, subjects will receive 12 weeks of treatment, after which there will be a 6-day taper period, during which subjects will reduce their dosage of topiramate gradually and then discontinue it completely. Daily reports during the treatment period will be obtained using interactive voice response (IVR) to identify subjective correlates of medication effects and to monitor medication use. Following the 12-week treatment period, subjects will be asked to return to the clinic for 3-month and 6-month post-treatment follow-up visits to evaluate the durability of treatment effects.

Two hundred men and women of European descent will be randomized to study medication. Subjects will be recruited using referrals from treatment programs throughout Philadelphia; IRB-approved advertisements on mass transit, on local radio and television stations and in newspapers, social media, and broadcast email messages at institutions that offer such a service and by posting/distributing recruitment materials in community and college settings. Respondents will initially be evaluated by telephone prior to an in-person visit to the Treatment Research Center of the University of Pennsylvania Perelman School of Medicine. The investigators will select subjects based on their genotype to ensure comparable numbers of individuals who are rs2832407*C-allele homozygotes and A-allele carriers. The investigators will block randomize subjects to balance the groups on treatment goal (i.e., reduced drinking or abstinence).

ELIGIBILITY:
Inclusion Criteria:

1. Determined to be physically healthy, based on medical history and physical examination and approval of the study physician
2. Age 18 to 70 years, inclusive
3. Self-identified European ancestry
4. Meets DSM-5 criteria for AUD
5. Average weekly ethanol consumption of >24 standard drinks for men and >18 standard drinks for women, with a weekly average of > 2 HDDs during the month before screening
6. Stated goal to reduce drinking to safe levels or to stop drinking
7. Able to read English at an 8th grade or higher level and no gross cognitive impairment
8. Willingness to nominate an individual who will know the subject's whereabouts to facilitate follow up during the study
9. Women of child-bearing potential (i.e., who have not had a hysterectomy, bilateral oophorectomy, tubal ligation or is less than two years postmenopausal): must be non-lactating and practicing a reliable method of birth control, and have a negative urine pregnancy test prior to the initiation of treatment. Examples of medically acceptable methods for this protocol include: the birth control pill, intrauterine device, injection of Depo-Provera, Norplant, contraceptive patch, contraceptive ring, double-barrier methods (such as condoms and diaphragm/spermicide), male partner sterilization, abstinence (and agreement to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence), and tubal ligation.
10. Willingness to provide signed, informed consent and commit to completing the procedures in the study

Exclusion Criteria:

1. A current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation, including direct bilirubin elevations of >110% or a transaminase elevation >300% of normal
2. A history of nephrolithiasis
3. A history of glaucoma
4. Current treatment with carbonic anhydrase inhibitors, due to the added risk of metabolic acidosis.
5. Current, serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe or psychotic major depression, panic disorder, borderline or antisocial personality disorder, organic mood or mental disorders, eating disorder, or imminent suicide or violence risk)
6. Current DSM-IV diagnosis of dependence on a drug other than alcohol or nicotine
7. A history of hypersensitivity to topiramate
8. Current regular treatment with a psychotropic medication (e.g., benzodiazepines, antidepressants), which affect neurotransmitter systems, or a medication to treat alcohol dependence
9. Currently taking any tricyclic antidepressant (e.g., Adapin (doxepin), Anafranil (clomipramine), Elavil (amitryptyline), Pamelor (nortryptyline), Tofranil (imipramine), Sinequan (doxepin)
10. Urine drug screen positive for recent use of opioids, cocaine, or amphetamines (may be repeated once and if the result is negative on repeat it is not exclusionary)
11. Because co-administration of topiramate with dolutegravir reduced plasma concentrations of the antiretroviral through induction of CYP3A, the use of dolutegravir is exclusionary.
12. Judged by the principal investigator or his designee to be an unsuitable candidate for receipt of an investigational drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry R Kranzler, M.D., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Kranzler HR, Feinn R, Pond T, Hartwell E, Gelernter J, Crist RC, Witkiewitz K. Post-treatment effects of topiramate on alcohol-related outcomes: A combined analysis of two placebo-controlled trials. Addict Biol. 2022 Mar;27(2):e13130. doi: 10.1111/adb.13130. PMID 35229945
- [Derived] Kranzler HR, Hartwell EE, Feinn R, Pond T, Witkiewitz K, Gelernter J, Crist RC. Combined analysis of the moderating effect of a GRIK1 polymorphism on the effects of topiramate for treating alcohol use disorder. Drug Alcohol Depend. 2021 Aug 1;225:108762. doi: 10.1016/j.drugalcdep.2021.108762. Epub 2021 May 21. PMID 34049101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from December 18, 2014 through August 1, 2019 at the University of Pennsylvania Treatment Research Center (Penn; n=164) and the Corporal Michael J. Crescenz Veterans Affairs Medical Center (CMCVAMC; n=6).
Pre-assignment Details: Participants completed an in-person visit, where they gave informed consent, underwent a medical history, physical examination, routine clinical laboratory testing, a urine drug screen, and, if appropriate, pregnancy testing. We excluded 150 participants based on the first in-person visit based on the inclusion/exclusion criteria from the protocol.
Groups:
- Topiramate + Medical Management: Topiramate 200 mg/day orally in two divided doses. Dose will be titrated upward over a six-week period, maintained for 6 weeks, then tapered over 6 days + Medical Management sessions for 15-25 minutes per study visit
  Medical Management: Medical Management (MM; Pettinati, 2004) will support subjects' efforts to reduce or stop their drinking.
- Placebo Pill + Medical Management: Inactive placebo with dosing schedule matched to intervention group + Medical Management sessions for 15-25 minutes per study visit
  Medical Management: Medical Management (MM; Pettinati, 2004) will support subjects' efforts to reduce or stop their drinking.
Period: Overall Study
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management
Started | 85 | 85
Completed | 66 | 71
Not Completed | 19 | 14
Not completed — Adverse medication effect | 11 | 2
Not completed — Lost to Follow-up | 6 | 5
Not completed — Personal time constraints | 2 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Relapse | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Customized [Mean (Standard Deviation); unit: years] | 52.3 (10.5) | 50 (12.8) | 51.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 61 | 60 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 85 | 85 | 170
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 85 | 85 | 170
Married or cohabiting [Count of Participants; unit: Participants] | 47 | 51 | 98
Genotype [Count of Participants; unit: Participants]
  CC genotype | 30 | 31 | 61
  AC/AA genotype | 55 | 54 | 109
Lifetime Major Depression [Count of Participants; unit: Participants] — Lifetime episode of Major depression based on DSM-IV (SCID-I/P)(First et al. 2001).
  Participants
    CC genotype | 7 | 11 | 18
    AC/AA genotype | 11 | 8 | 19
Lifetime Anxiety Disorder [Count of Participants; unit: Participants] — Lifetime episode of Anxiety based on DSM-IV (SCID-I/P)(First et al. 2001).
  Participants
    CC genotype | 5 | 4 | 9
    AC/AA genotype | 6 | 19 | 25
Drinking Days 90days prior to screening [Mean (Standard Deviation); unit: Drinking days] — Drinking day measured in standard drinks.
  Drinking days | 87.2 (16.5) | 86.3 (16.8) | 86.5 (17.01)
Heavy drink days 90 days prior to screening [Mean (Standard Deviation); unit: Heavy drinking days] — Heavy drinking day measured as 5 or greater standard drinks for men and 4 or greater standard drinks for women in a day.
  Heavy drinking days | 73.8 (23.5) | 68.7 (25.6) | 68.9 (26.58)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Heavy Drinking Days by Medication Group (Timeline Follow Back Calendar).
Description: The number of Heavy Drinking Days during 12 weeks of treatment in the topiramate and placebo groups.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Heavy drinking days
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management
Number analyzed (Participants) | 85 | 85
Heavy drinking days | 29.00 (23.82) | 41.25 (26.38)

2. Primary Outcome: Frequency of Heavy Drinking Days Per Day by Medication and Genotype Group (Timeline Follow Back Calendar).
Description: Number of Heavy Drinking Days in the last week of the 12 week treatment phase by medication group and rs2832407 genotype group.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Heavy drinking days during week 12
Groups:
- Genotype CC Topiramate + Medical Management: Topiramate 200 mg/day orally in two divided doses. Dose will be titrated upward over a six-week period, maintained for 6 weeks, then tapered over 6 days + Medical Management sessions for 15-25 minutes per study visit
  Medical Management: Medical Management (MM; Pettinati, 2004) will support subjects' efforts to reduce or stop their drinking.
- Genotype CC Placebo Pill + Medical Management; Genotype AA/AC Placebo Pill + Medical Management: Inactive placebo with dosing schedule matched to intervention group + Medical Management sessions for 15-25 minutes per study visit
  Medical Management: Medical Management (MM; Pettinati, 2004) will support subjects' efforts to reduce or stop their drinking.
- Genotype AA/AC Topiramate + Medical Management: opiramate 200 mg/day orally in two divided doses. Dose will be titrated upward over a six-week period, maintained for 6 weeks, then tapered over 6 days + Medical Management sessions for 15-25 minutes per study visit
  Medical Management: Medical Management (MM; Pettinati, 2004) will support subjects' efforts to reduce or stop their drinking.
Arm/Group | Genotype CC Topiramate + Medical Management | Genotype CC Placebo Pill + Medical Management | Genotype AA/AC Topiramate + Medical Management | Genotype AA/AC Placebo Pill + Medical Management
Number analyzed (Participants) | 30 | 31 | 55 | 54
Heavy drinking days during week 12 | 1.86 (2.27) | 3.17 (2.69) | 2.24 (2.46) | 3.14 (2.68)

3. Primary Outcome: Numbers of Drinking Days Over 12 Weeks Treatment by Medication Group.
Description: Numbers of drinking days over 12 week treatment phase by medication group. Data was collected using timeline follow back calendar.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Drinking days
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management
Number analyzed (Participants) | 85 | 85
Drinking days | 58.58 (25.35) | 65.14 (22.31)

4. Other Pre Specified Outcome: Adverse Effects in Study Participants (Questionnaire)
Description: Cumulative number of adverse events as assessed at each study visit to determine the safety of topiramate.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Number of adverse events
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management
Number analyzed (Participants) | 85 | 85
Number of adverse events | 3.5 (1.7) | 2.6 (1.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Frequency, type, and severity of adverse effects will be assessed at each study visit to determine the safety of topiramate.
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management
All-Cause Mortality (participants affected / at risk) | 1/85 | 1/85
Serious Adverse Events (participants affected / at risk) | 1/85 | 1/85
Other Adverse Events (participants affected / at risk) | 80/85 | 76/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate + Medical Management (N=85) | Placebo Pill + Medical Management (N=85)
exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
alcohol-related relapse (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate + Medical Management (N=85) | Placebo Pill + Medical Management (N=85)
Paresthesia (General disorders) | 46 | 9
Headache (General disorders) | 21 | 15
Dysgeusia (General disorders) | 30 | 5
Pain and discomfort (General disorders) | 16 | 17
Fatigue (General disorders) | 21 | 10
Upper respiratory infections (General disorders) | 21 | 10
Eye Disorders (General disorders) | 17 | 7
Speech/Language abnormalities (General disorders) | 18 | 3
Insomnia (General disorders) | 12 | 8
Somnolence (General disorders) | 12 | 6
Diarrhea (General disorders) | 8 | 9
Injuries NEC (General disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02371889/Prot_SAP_002.pdf
  • Informed Consent Form (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02371889/ICF_003.pdf